CLINICAL TRIAL: NCT05595863
Title: Single Photon Emission Computed Tomography/Computed Tomography With Pentavalent 99mTc Dimercaptosuccinic Acid in Patients With Brain Glioma; Correlation With IDH Mutation
Brief Title: Correlation Between SPECT/CT and IDH Mutation in Brain Glioma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Radwa Gaber Elsaady, researcher, Assiut University
Other Study IDs: 123glioma
Record Dates: First submitted 2022-10-23; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Brain Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Major advances in cancer genetics over the past decade have revealed that the genes encoding IDHs are frequently mutated in a variety of human malignancies, including gliomas.Pentavalent 99mTc dimercaptosuccinic acid (99mTc (V) DMSA), is a nonspecific tumor targeting SPECT radiotracer, that has been used for imaging of various tumors including lung and breast carcinoma. However, to date, scarce reports discussed the utility of DMSA-V in patients with glioma.SPECT has the advantages of being widely available and not expensive. Multiple SPECT tracers have been explored. Of them Thallium-201 and 99 mTc-MIBI are, possibly, the most extensively discussed.

DETAILED DESCRIPTION:
Every year, nearly100,000 people worldwide are diagnosed as having brain gliomas. Although it comprises <1% of all newly diagnosed cancers, brain glioma is associated with substantial mortality and morbidity. Gliomas are intrinsic brain tumors that originate from neuroglial progenitor cells. Conventional therapies, including surgery, chemotherapy, and radiotherapy, have achieved limited improvements in the prognosis of glioma patients.

Radiation therapy to the brain may lead to postradiation injury which typically occurs within the first 3 to 12 months after radiotherapy but it was reported up to several years and even decades later. The clinical picture of radiation necrosis (RN) is variable and may include seizures, headache, personality changes, and neurologic deficits. These symptoms mimic tumor recurrence and differentiation between the two entities clinically or even by conventional radiological modalities is difficult but is necessary because the two conditions have different treatment modalities and prognosis.

SPECT has the advantages of being widely available and not expensive. Multiple SPECT tracers have been explored. Of them Thallium-201 and 99 mTc-MIBI are, possibly, the most extensively discussed. The main disadvantage of 201Tl is the lower spatial resolution, relatively large radiation dose, and the reported high false positive results. Normal uptake of MIBI in the choroid plexus may be confounding for assessing tumors around the ventricles.

Pentavalent 99mTc dimercaptosuccinic acid (99mTc (V) DMSA), is a nonspecific tumor targeting SPECT radiotracer, that has been used for imaging of various tumors including lung and breast carcinoma. However, to date, scarce reports discussed the utility of DMSA-V in patients with glioma.

Isocitrate dehydrogenase (IDH) enzymes, of which there are three isoforms, are essential enzymes that participate in several major metabolic processes, such as the Krebs cycle, glutamine metabolism, lipogenesis and redox regulation.

Major advances in cancer genetics over the past decade have revealed that the genes encoding IDHs are frequently mutated in a variety of human malignancies, including gliomas, acute myeloid leukaemia, cholangiocarcinoma, chondrosarcoma and thyroid carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pathologically proven glioma.
* patients conscious to provide informed consent.

Exclusion Criteria:

* Pregnant women.
* severely ill patients and those with disturbed conscious level,
* patients who were judged that they cannot lie down comfortably without movement for at least 20 min..

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Glioma patients visiting the nuclear medicine unit in Assiut university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
degree of 99mTc-DMSA (V) uptake at SPECT/CT. | Baseline
  measured by calculating quantitative index of 99m Tc-DMSA (V) uptake by SPECT/CT as a biomarker for IDH mutation

SECONDARY OUTCOMES:
IDH mutation | Baseline
  measured by immunohistochemistry technique using the anti-IDH antibody

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31227792/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21912937/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/20143189/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7250901/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15586883/